CLINICAL TRIAL: NCT01400321
Title: PEERS Multicenter OsseoSpeedTM TX Profile Implant: German Astra Soft Tissue (GAST) Maintenance Study An Open, Prospective Observational Study to Evaluate Implant Stability, Marginal Bone and Soft Tissue Maintenance of the Astra Tech Dental Implant System: OsseoSpeedTM TX Profile Implant in Patients With Tooth Loss in the Aesthetic Zone or the Posterior Atrophied Mandible
Brief Title: PEERS Multicenter Osseospeed TM TX Profile Implant: German Astra Soft Tissue (GAST) Maintenance Study
Acronym: GAST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Dr. Wilfried Wagner, Prof. Dr. Dr. Wilfried Wagner, Johannes Gutenberg University Mainz
Other Study IDs: GAST
Record Dates: First submitted 2011-06-07; First posted 2011-07-22 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Inclined Atrophy of the Distal Mandible; Socket Like Atrophy of the Aesthetic Zone
Keywords: dental implant; soft tissue maintenance; bone remodelling; inclined atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Distal region: Patients with loss of tooth in the premolar and molar region of the atrophied mandible
- aesthetic zone: Patients with loss of tooth within the aesthetic zone (canine to canine)

SUMMARY:
The open, prospective, non-controlled observational study is designed to provide information on the short-, medium- and long-term clinical performance of the Astra Tech OsseospeedTM implant surface in combination with a special implant design. The study will provide information on implant survival and soft tissue and bone maintenance as clinical performance of the OsseoSpeedTM TX Profile Implant in the aesthetic zone or the posterior mandible with socket like atrophy.

DETAILED DESCRIPTION:
Within the new OsseoSpeedTM TX Profile Implant from Astra Tech a special surface modification treated with diluted hydrofluoric acid is combined with an inclined implant-abutment interface to support soft tissue and marginal bone maintenance in the aesthetic zone or the socket like atrophy in the mandible. Pre-clinical studies of the OsseospeedTM modification support improvement in osseointegration. Both aspects are of special clinical interest in critical situations e.g. reduced bone quantity and quality or in case of socket atrophy with loss of the papillae. The outcome variables of interest are implant survival and the marginal bone and soft tissue response for clinical evaluation of the OsseoSpeedTM TX Profile Implant from Astra Tech. In contrast to the original treatment protocol with a healing period of 3 and 6 months for maxilla and mandible, respectively, the healing period is reduced to 3 months following the recent literature with equal clinical results. Within the present study implants will heal in a transgingival mode and loaded after a healing period of 3 months. For special indications in the aesthetic zone the implants may optionally be loaded following an early loading protocol, which comprehend temporary loading within 48h after implant insertion. Overall implant survival rates are high. However, for implants placed immediately after tooth extraction in the esthetic zone or in the socket like atrophied mandible survival rates are lower. The special physiology of bone resorption in the aesthetic zone exhibit high requirements for soft tissue and bone maintenance for good clinical long term results. Differences in pattern of marginal bone response have been described for different implant systems. The extend of bone loss as also the pattern of remodeling as reaction to OsseospeedTM surface and the special shape of the OsseoSpeedTM TX Profile Implant will be investigated within the present study.

ELIGIBILITY:
Inclusion Criteria:

* loss of tooth aesthetic zone (a maximum of 4 implants)
* loss of tooth at the distal mandible (distal canine) (a maximum of 4 implants)
* presence of inclined alveolar ridge profile
* antagonists are natural teeth or fixed prosthesis

Exclusion Criteria:

* < 18 years
* Tumour or irradiation
* bisphosphonate or cortisone intake
* Diabetes mellitus
* Mental illness or disorder with affection of compliance
* Consumption of > 20 cigarettes/day
* Bruxism
* Acute Mucosal infection or illness (e.g. acute Parodontitis, Pemphigus, Lichen)
* Relation of Crown to Implant ratio of > 1
* No clinical primary stability of the implant after insertion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with tooth loss in the aesthetic zone or in the distal mandible with socket like atrophy. The antagonists should be natural teeth or a fixed prosthesis.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Implant survival | after 24 months
  How many implants are in situ after an observational period of 24 months (2 years). Data presentation will be a Kaplan Meier Estimate.

SECONDARY OUTCOMES:
Marginal bone adaption | after 24 months
  Marginal bone adaptation will be assessed clinically as probing depth on the lingual aspect of insertion. In addition marginal bone adaption will be followed as the distance from the implant reference point to the most coronal bone-to-implant contact on the mesial and distal side of the implant on intraoral radiographs with paralleling technique. Periapical radiographs will be taken pre- and postoperatively at 24 months follow-up visit. A change in marginal bone will be recorded as positive or negative shift compared to the baseline (preoperatively measured bone height).
Pinc aesthetic parameter | after 24 months
  Pinc aesthetic score evaluation as previously described by Fürhauser and measurement of width of keratinized mucosa and clinical crone length. Data evaluation will be a negative or positive shift compared to the preoperatively evaluated data.
periodontal parameter | after 24 months
  Clinical evaluation of of probing depth in mm (mesial, distal, oral and vestibular), bleeding on probing and Plaque Index as described by Sillness and Löe. Data evaluation will be a negative or positive shift compared to the preoperatively evaluated data.
Detection and description of implant related complications and other adverse and serious adverse events | over the study period (24 months)
  Complications are characterized by any failure (mechanical or other) of the implant and/or the prosthetic restoration, as well as the treatment of such failures and will be recorded. The following complications must be reported to the Principal Investigator within 4 working days:
  * Failed osseointegration
  * Lost osseointegration
  * Fixture fracture Adverse events and serious adverse events detection and reporting following GCP-ICH

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried Wagner, MD, DMD, PHD, Principal Investigator — Department of Oral and Maxillofacial Surgery, University Mainz, Medical Center
Locations (28):
- Germany (28):
  - Department of Oral and Maxillofacial Surgery, University Mainz, Medical Center, Mainz, Rhineland-Palatinate
  - MSc. E. Trilck, Berlin
  - Dr.Dr. U. Schwarzott, Berlin
  - Dr. M. Loeck, Berlin
  - Dr. G. Körner, Bielefeld
  - PD.Dr.Dr. E. Keese, Braunschweig
  - Klinik für MKG Chirurgie Dortmund, Dortmund
  - Dr.Dr. V. Michalczik, Essen
  - Dr. M.Sc. Gau, Euskirchen
  - Dr. M. Schlee, Forchheim
  - Dr. Borrmann, Freiberg
  - Dr. H. Steveling, Gernsbach
  - Dr. Dr. St. Kahnel, Hamburg
  - Dr. U. Konter, Hamburg
  - K. Bothe, Hanover
  - Klinik für MKG Chirurgie MH Hannover, Hanover
  - Dr. Ch. Mertens, Heidelberg
  - Dr. W. Knöfler, Leipzig
  - Dr. R. Noelken, Lindau
  - Dr.Dr. R. Wörtche, Lorsch
  - Dr. Dr. Barth, Mannheim
  - Dr. P. Rauch, Melsungen
  - Dr. MMsc Dirlewanger, Nagold
  - Prof. Dr. H. Visser, Oldenburg
  - Dr.Dr. M. Kestel, Rückersdorf
  - Dr. J. U. Wiegner, Saalfeld
  - Dr. M. Riedl, Stein
  - Tagesklinik für Kiefer- und Plastische Gesichtschirurgie, Wiesbaden

REFERENCES:
- [Derived] Schiegnitz E, Noelken R, Moergel M, Berres M, Wagner W. Survival and tissue maintenance of an implant with a sloped configurated shoulder in the posterior mandible-a prospective multicenter study. Clin Oral Implants Res. 2017 Jun;28(6):721-726. doi: 10.1111/clr.12869. Epub 2016 May 13. PMID 27172991